CLINICAL TRIAL: NCT05115552
Title: Comparison Between Urocortin 2 and Brain Type Natriuretic Peptide as a Biomarker in Patients With Acute Heart Failure
Brief Title: Comparison Between Urocortin 2 and Brain Type Natriuretic Peptide
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christen Saad Welliam, resident, Assiut University
Other Study IDs: Urocortin 2 Biomarker
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Urocortin 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Evaluation of the role of serum urocortin 2 levels in acute decompensated HF patients and their association with clinical and echocardiographic findings.
2. Assessment of the clinical utility of urocortin 2 in monitoring AHF patients.
3. Comparison between urocortin 2 and BNP as a biomarker in AHF patients

DETAILED DESCRIPTION:
Heart failure (HF) is a clinical syndrome with symptoms and/or signs caused by a structural and/ or functional cardiac abnormality and corroborated by elevated natriuretic peptide levels and/or objective evidence of pulmonary or systemic congestion. (1) .The pathophysiology of HF is a complex interplay of genetic and multiple molecular mechanisms (from inﬂammation to hormonal pathways) performing in the composite network of the cardiovascular system environment. (2).

Monitoring of biomarkers in HF can be used to make an initial diagnosis, to aid in prognostic stratification, and to identify a patient's response to therapeutic intervention. (3).

Natriuretic peptide (NP) concentrations are quantitative plasma biomarkers for the presence and severity of haemo-dynamic cardiac stress and heart failure. (4). That facilitate renal filtration and sodium excretion whilst suppressing the vasoconstrictor sodium, retaining Renin angiotensin aldosterone system and exerting a tonic anti-trophic effect. (5). But the natriuretic peptide levels are significantly affected by weight, the NT- proBNP in obese subjects is much lower than normal weight subjects. (6). Other factors that affect BNP levels including gender, age and renal disease

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acute decompensated heart failure.

Exclusion Criteria:

* Acute coronary syndrome or stroke in the past 3 months.
* Severe chronic kidney disease.
* Severe valve disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: both gender above 18 years old with acute decompensated heart failure without ACS or stroke in the past 3 months or severe valvular disease or severe CKD .
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the role of serum urocortin 2 levels | baseline
  Evaluation of the role of serum urocortin 2 levels in acute decompensated HF patients and their association with clinical and echocardiographic findings.
Assessment of the clinical utility of urocortin 2 in monitoring AHF patients | baseline

SECONDARY OUTCOMES:
Comparison between urocortin 2 and BNP | baseline
  Comparison between urocortin 2 and BNP as a biomarker in AHF patients(which is more specific for AHF patients )